CLINICAL TRIAL: NCT01417611
Title: The Usefulness of I-scan in Screening Colonoscopy: A Randomized Controlled Trial
Brief Title: The Usefulness of I-scan in Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Hospital (Other)
Responsible Party: Sung Noh Hong, M.D., Digestive Disease Center, Healthcare Center, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KUMCHSN02
Record Dates: First submitted 2010-07-27; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Colorectal Neoplasm
Keywords: screening colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- i-scan-CE/SE (Experimental): Study Group using i-scan SE and CE mode: i-scan-CE/SE group was explored whole colon from the cecum to the rectum with i-scan-CE 2+ and SE 2+ mode. They had a chance to switch from i-scan to WL to perform polyp removal using cold biopsy or polypectomy
  Interventions: Procedure: i-scan CE, SE, TE mode
- i-scan-CE/SE/TE-c (Experimental): Study Group using i-scan SE & CE mode as well as TE-c mode: i-scan-CE/SE/TE-c group was explored whole colon from the cecum to the rectum with i-scan CE2+, SE2+, TE-c mode. They had a chance to switch from i-scan to WL to perform polyp removal using cold biopsy or polypectomy
  Interventions: Procedure: i-scan CE, SE, TE mode

INTERVENTIONS:
Procedure: i-scan CE, SE, TE mode — I-scan technology is the newly developed image enhanced endoscopy technology, classified as a digital contrast method among endoscopic imaging techniques. I-scan has three modes of image enhancement, i.e. surface enhancement (SE); contrast enhancement (CE); and tone enhancement (TE). The three modes (SE, CE and TE) are arranged in series, therefore, it is possible to apply two or more of these three modes at one time. Switching the levels or modes of enhancements can be done on a real-time basis, without any time lag by pushing a relevant button, thus enabling efficient endoscopic observation.
  Other Names: EPKi

SUMMARY:
Image-enhanced endoscopy in screening colonoscopy

1. useful tool for detecting subtle epithelial lesions
2. useful tool for predicting real-time histology of epithelial lesions. Among image-enhancing techniques, i-SCAN is new developed and the practical usefulness of i-scan for screening colonoscopy has not been investigated yet.

DETAILED DESCRIPTION:
New technologies have been developed to enhance the visualization of colorectal mucosa to unmask even minute mucosal lesions and identify neoplastic lesion from non-neoplastic lesions. In particular, there appears to be strong evidence that pan-colonic chromoendoscopy enhances the detection of colorectal neoplasm in the colon and rectum. However, this technique is time-consuming because of both the dye spraying and suction of collected dye in the dependent portion, and therefore it is unsuitable for routine application. To overcome this inconvenience, optical-digital method involves conversion of the optical characteristics of the light used for illumination or imaging with a light source differing in optical characteristics from ordinary white light (WL), such as narrow band imaging (NBI), Fujinon imaging color enhancement (FICE), auto-fluorescence imaging (AFI) and infra-red imaging (IRI).

I-scan technology is the newly developed image enhanced endoscopy technology, classified as a digital contrast method among endoscopic imaging techniques.19 I-scan has three modes of image enhancement, i.e. surface enhancement (SE); contrast enhancement (CE); and tone enhancement (TE). The three modes (SE, CE and TE) are arranged in series, therefore, it is possible to apply two or more of these three modes at one time. Switching the levels or modes of enhancements can be done on a real-time basis, without any time lag by pushing a relevant button, thus enabling efficient endoscopic observation. Furthermore, while NBI) images are much darker than conventional white light (WL) images, i-scan images are as bright as conventional WL images, therefore, i-scan is able to observe much larger areas in a distant view compared with NBI. Consequently, i-scan might be more useful for performing screening endoscopy).

However, the actual usefulness of I-scan in enhancing the detection of colonic neoplastic lesions is not known yet in screening colonoscopy. Therefore, we tried to evaluate the hypothesis that, in subjects undergoing colonoscopy screening, the routine application of i-scan during withdrawal could improve adenoma detection as compared with standard WL examination.

ELIGIBILITY:
Inclusion Criteria:

* a consecutive series of asymptomatic average-risk subjects aged 40-75 years who underwent first screening colonoscopy at the Healthcare Center of Konkuk University Medical Center in Seoul, Korea

Exclusion Criteria:

* (i) the colonoscopy did not reach the cecum, (ii) the bowel preparation was poor or inadequate (iii) patients taking anticoagulants that precluded removal of polyps during colonoscopy, (iv) patients had a history of bowel resection, or (v) patients who refused to participate or were unable to provide informed consent to the study (vi) patients with melanosis coli

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
polyp/adenoma detection rate (per-polyp/adenoma analysis and per-patient analysis) | up to 24 weeks
  To compare the polyp/adenoma detection rate (per-polyp/adenoma analysis and per-patient analysis) among conventional WL, i-scan-CE/SE or i-scan-CE/SE/TE-c groups.

SECONDARY OUTCOMES:
characterization of polyp | up to 24 weeks
  To differentiate the adenomatous polyp from non-adenomatous polyp using colonoscopic finding

CONTACTS AND LOCATIONS:
Overall Officials: Sung Noh Hong, M.D., Principal Investigator — Konkuk University Medical Center
Locations (1):
- Healthcare Center, Digestive Disease Center, Konkuk University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong SN, Choe WH, Lee JH, Kim SI, Kim JH, Lee TY, Kim JH, Lee SY, Cheon YK, Sung IK, Park HS, Shim CS. Prospective, randomized, back-to-back trial evaluating the usefulness of i-SCAN in screening colonoscopy. Gastrointest Endosc. 2012 May;75(5):1011-1021.e2. doi: 10.1016/j.gie.2011.11.040. Epub 2012 Feb 28. PMID 22381530